CLINICAL TRIAL: NCT04219592
Title: Comparing IgG-4 Levels in Systemic Sclerosis Patients vs. Healthy Controls
Brief Title: IgG-4 Levels in Systemic Sclerosis
Acronym: SSc-IgG4
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Noa Rabinowicz, Principal investigator, Meir Medical Center
Other Study IDs: MMC-110-19
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Systemic Sclerosis
Keywords: SSc; IgG4
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — sera from healthy participants purchased from MDA will be used as control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SSc: 74 SSc patients aged 18 - 85
  Interventions: Diagnostic Test: IgG4 measurement (non-interventional, just obtaining data from medical records)
- Healthy controls: 80 Healthy blood-donors aged 18 - 85
  Interventions: Diagnostic Test: IgG4 measurement (non-interventional, just obtaining data from medical records)

INTERVENTIONS:
Diagnostic Test: IgG4 measurement (non-interventional, just obtaining data from medical records) — IgG4 measurement in mg/dL

SUMMARY:
This is an observational - non interventional study. The investigators will compare IgG4 levels of 80 healthy donors (from Israel blood bank - MDA) and 80 Systemic Sclerosis patients from Meir Medical Center.

DETAILED DESCRIPTION:
IgG4 levels will be obtained from medical records of 80 SSc patients between the years 2000-2019. These will be compared to IgG4 levels from sera of 80 healthy donors (from Israel blood-bank - MDA). Correlations between IgG4 levels and the following will be made: age, sex, disease type (limited or diffused SSc), disease duration, medications.

ELIGIBILITY:
Inclusion Criteria:

* SSc patients

Exclusion Criteria:

* other chronic co-morbidities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical records of SSc patients from Meir Medical Center
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
IgG4 measurement | 4 months
  quantifying IgG4 in each group and in SSc subgroups based on disease type, organs involved, medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No
not relevant